CLINICAL TRIAL: NCT03526679
Title: A Single-arm Phase Ib/II Study of the Combination of Lenvatinib and Eribulin in Advanced Adipocytic Sarcoma and Leiomyosarcoma (LEADER Study)
Brief Title: Lenvatinib and Eribulin in Advanced Soft Tissue Sarcoma
Acronym: LEADER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201801101MIPB
Record Dates: First submitted 2018-04-19; First posted 2018-05-16 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Leiomyosarcoma; Liposarcoma; Soft Tissue Sarcoma Adult; Advanced Cancer
Keywords: soft tissue sarcoma; phase Ib/II; advanced cancer
MeSH Terms: conditions — Leiomyosarcoma; Liposarcoma; Sarcoma | interventions — eribulin; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): The combination of lenvatinib and eribulin
  Interventions: Drug: Eribulin; Drug: Lenvatinib

INTERVENTIONS:
Drug: Eribulin — lenvatinib 14mg po daily; eribulin 1.1mg/m2 D1, D8, every 21 days
  Other Names: Halaven
Drug: Lenvatinib — lenvatinib 14mg po daily; eribulin 1.1mg/m2 D1, D8, every 21 days
  Other Names: Lenvima

SUMMARY:
This study is designed to test the safety and efficacy of the combination of lenvatinib, a drug that can inhibit the growth of supplying vessels around the tumors, and eribulin, a chemotherapy drug that targets the cancer cell during mitosis, in inoperable or metastatic adipocytic sarcoma and leiomyosarcoma.

DETAILED DESCRIPTION:
Recently, the US Food and Drug Administration (FDA) granted approval to eribulin for the treatment of adipocytic sarcoma who have received a prior anthracycline-containing regimen based on a Phase III study results of improved overall survival (OS) as compared with the standard treatment dacarbazine. In the leiomyosarcoma cohort of the study, although eribulin did not demonstrate a significant benefit over dacarbazine, still about 5.1% of leiomyosarcoma patients treated with eribulin had a partial response, suggesting that eribulin may have activity against leiomyosarcoma. However, the overall response rate (ORR) and progression-free survival (PFS) remained unsatisfactory in the two most common soft tissue sarcoma (STS) subtypes-adipocytic sarcoma and leiomyosarcoma, prompting new therapeutic options of STS patients.

Anti-angiogenic therapies had shown promising results in soft tissue sarcoma (ST). Pazopanib, an anti-angiogenic multi-kinase inhibitor, has shown clinical benefit with a longer median PFS of 4.6 months versus placebo in STS patients refractory to at least one line of systemic chemotherapy. Another anti-angiogenic targeted therapy, regorafenib, showed significant improvement in PFS as compared with placebo in various STS. In a phase I study of lenvatinib for solid tumors in Japan, 4 out of 6 leiomyosarcoma patients has tumor decreased more than 10%. Moreover, other tyrosine receptor targets of lenvatinib, such as fibroblast growth factor receptor (FGFR) and platelet-derived growth factor receptor (PDGFR), may also plays a role in treating STS. In high-grade STS patients, about 30% of patients had FGFR1 amplification or overexpression. FGFR1-overexpression STS cell lines are sensitive to FGFR inhibitors such as BGJ398 and AZD45475. Furthermore, a monoclonal antibody of PDGFR alpha, olaratumab, was recently approved by the FDA in combination with doxorubicin for advanced STS based on a median 10-month OS benefit compared to doxorubicin only in a randomized phase II trial.

It has been demonstrated in various cancer types that an increased quantity of tumor infiltrating lymphocyte (TILs) is associated with increased response to chemotherapy or improved prognosis. One of the factors that had been shown to impede the migration and trafficking of TILs into tumor is vascular endothelial growth factor (VEGF). In renal cell carcinoma, treatment with bevacizumab, an anti-VEGF antibody, or in combination with atezolizumab, increased the recognition of tumor antigen, increased expression of major histocompatibility complex (MHC) class I receptor on tumor cells, and the amount of TIL migration into the tumor stroma9. Many of the STS were detected with scarce TILs in the tumor microenvironment, thus it would be interesting to see if anti-angiogenic tyrosine kinase inhibitors could adjust the tumor microenvironment toward a more chemotherapy-friendly milieu.

Thus, we would like to propose a clinical trial to understand the anti-tumor activity of the combination of lenvatinib and eribulin in advanced STS patients.

ELIGIBILITY:
Inclusion criteria

1. A histological confirmed adipocytic sarcoma (dedifferentiated, myxoid, or pleomorphic) or leiomyosarcoma that is either inoperable locally advanced or metastatic
2. Advanced adipocytic sarcoma and leiomyosarcoma who have received no more than 2 lines of systemic chemotherapy in the advanced setting (not including adjuvant chemotherapy).
3. At least one measurable tumor according to RECIST 1.1. If the measurable lesion has previously received radiotherapy, the tumor must be a progressive lesion after radiotherapy.
4. ECOG PS 0 or 1 or Karnofsky performance status (KPS) ≥ 70
5. Patients must have adequate organ function and marrow reserve measured within 14 days prior to randomization as defined below:

   * Hemoglobin ≥ 9.0 g/dL;
   * Absolute neutrophil count ≥ 1,500 /µL;
   * Platelets ≥ 75,000/µL;
   * Total bilirubin ≤ 1.5 x upper normal limit;
   * aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) ≤ 2.5 x upper normal limit; for patients with liver metastases AST(SGOT)/ALT(SGPT) ≤ 5 x upper normal limit is allowed;
   * Serum creatinine ≤ 1.5mg/dL or creatinine clearance ≥ 50ml/min;
   * activated partial thromboplastin time (aPTT) < 1.5 x upper normal limit (unless on therapeutic anti-coagulation);
   * Proteinuria ≤ 1+ with urine dipstick, if > 1+, 24-hour urine protein must be ≤ 1 g
6. Age 20 or older.
7. Patient's life expectancy is more than 3 months
8. All women of childbearing potential must have a negative pregnancy test obtained within 72 hours before starting therapy.
9. Patients with reproductive potential must use effective contraception (hormone or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after the completion of therapy.
10. Patient needs to have adequate wash-out period from previous systemic treatment(s):

(1) 2 weeks for any other oral anti-cancer targeted agents (2) 3 weeks for any other cytotoxic chemotherapy (except for mitomycin-C, which will require 6 weeks) (3) 3 weeks for monoclonal antibodies, including immune checkpoint inhibitors

Exclusion criteria

1. Patients who had received lenvatinib or eribulin treatment
2. Patients who had leptomeningeal metastasis, either diagnosed by brain imaging study or confirmed by cerebrospinal fluid cytology examination (patients with brain metastasis that are under control is eligible).
3. Patients with clinical signs or symptoms of gastrointestinal obstruction and who require parenteral hydration and/or nutrition because of obstruction.
4. Patients with uncontrollable hypertension (defined as systolic blood pressure over 140mmHg and/or diastolic pressure over 90mmHg despite anti-hypertensive medications)
5. Patients with the following cardiac disease

   * Prolongation of corrected QT (QTc) interval to >480 milliseconds (ms).
   * Significant cardiovascular impairment: history of (a) congestive heart failure greater than New York Heart Association (NYHA) Class II; (b) unstable angina; (c) myocardial infarction; (d) stroke; or (e) cardiac arrhythmia associated with hemodynamic instability within 6 months of the first dose of study drugs.
6. Bleeding subjects at risk for severe hemorrhage.
7. Arterial thromboembolic event within the past 6 months, including transient ischemic attack, cerebrovascular accident, unstable angina, or myocardial infarction.
8. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment.
9. History of allergic reaction to compounds of similar chemical composition to the study drugs
10. Pregnancy or lactation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2025-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Wu Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei, Taiwan
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Derived] Chen TW, Hsu CL, Hong RL, Lee JC, Chang K, Yu CW, Chen SC, Guo JC, Chen ML, Hsu MC, Kung TF, Cheng AL, Yen CC. A Single-Arm Phase Ib/II Study of Lenvatinib plus Eribulin in Advanced Liposarcoma and Leiomyosarcoma. Clin Cancer Res. 2022 Dec 1;28(23):5058-5065. doi: 10.1158/1078-0432.CCR-22-2092. PMID 36129471

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental arm
Started | 30
Completed | 28
Not Completed | 2
Not completed — still under treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 59 [29 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 30
Region of Enrollment [Number; unit: participants]
  Taiwan | 30

OUTCOME MEASURES:

1. Primary Outcome: The Objective Response Rate (ORR) Based on RECIST 1.1
Description: We will measure the radiographic changes of the tumor based on a prespecified criteria called RECIST (Response evaluation criteria in solid tumors). A tumor decreased in the sum of longest diameters of measurable tumors of more than 30% is considered responsive; a growth of tumor more than 20% in the sum of the longest diameter is considered disease progression; and shrinkage or growth between these intervals is considered stable disease (SD).
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental arm
Number analyzed (Participants) | 30
Participants | 6

2. Secondary Outcome: The Proportion of Patients Who Are Progression-free and Alive at 24 Weeks
Description: We will measure how many patients (proportion) of the participants that the tumor has progressed in the first 24 weeks of treatment
Time Frame: 24 weeks
Population: IIT population
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental arm
Number analyzed (Participants) | 30
Participants | 30

3. Secondary Outcome: Overall Survival (OS) Rate at 12-months
Description: The definition of 12-months OS rate is the percentage of patients who had NOT has an event before or at 12 months. An event is defined as follows: Death due to any cause.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-01

4. Secondary Outcome: Overall Survival (OS) Rate at 6 Months
Description: The definition of 6 months OS rate is the percentage of patients who had NOT has an event before or at 6 months. An event is defined as follows: Death due to any cause.
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Toxicities will be assessed according to CTCAE 4.03. The number of all grade toxicities will be recorded
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 years
Arm/Group | Experimental arm
All-Cause Mortality (participants affected / at risk) | 12/30
Serious Adverse Events (participants affected / at risk) | 20/30
Other Adverse Events (participants affected / at risk) | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental arm (N=30)
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 4
neutrophil decrease (Blood and lymphatic system disorders) | 11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental arm (N=30)
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT03526679/Prot_SAP_000.pdf